CLINICAL TRIAL: NCT01525576
Title: Efficacy of an Internet-based Booster Program for Obsessive-compulsive Disorder: A Randomized Controlled Trial
Brief Title: Booster as an Adjunct to Internet-based Cognitive Behavior Therapy (CBT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Christian Rück, Dr Christian Ruck, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OCD_B
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Obsessive-compulsive Disorder
Keywords: booster program; internet; cbt; Study the specific effects of adding a booster program
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Color Vision Defects | interventions — Immunization, Secondary

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): No offer of booster program.
- Booster (Experimental): 3 week booster program + 2 additional weeks two months later for follow-up.
  Interventions: Behavioral: Booster

INTERVENTIONS:
Behavioral: Booster — 3 week booster program + 2 additional weeks two months later for follow-up.
  Arms: Booster

SUMMARY:
In this trial, we test if adding an Internet-based booster program to regular Internet-based cognitive behavior therapy (ICBT) is effective for patients with obsessive-compulsive disorder (OCD).

DETAILED DESCRIPTION:
Written consent form. Completing ICBT in our previous study: Please see NCT01347099 for more details.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent
* Previously enrolled in our randomized controlled trial testing ICBT for OCD: NCT01347099

Exclusion Criteria:

* Suicidal ideation that could jeopardize participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of obsessions and compulsions after 3, 8 and 20 months after baseline. | 3 months before treatment, 3 weeks after treatment starts, 6 and 18 months after treatment has ended
  Yale Brown Obsessive Compulsive Scale (Y-BOCS). Analysis will examine the frequency of relapse from remission between the groups. Furthermore, frequency of incremental cases of remission will be compared between the groups.

SECONDARY OUTCOMES:
Change from Baseline of obsessions and compulsions after 8 and 20 months. | 3 months before treatment, 6 and 18 months after treatment has ended
  Obsessive Compulsive Scale - Revised (OCI-R)
Change from Baseline of obsessions and compulsions after 8 and 20 months. | 3 months before treatment, 6 and 18 months after treatment has ended
  Trimbos Institute Cost-assessment for Psychiatry (TIC-P)
Change from Baseline of obsessions and compulsions after 8 and 20 months. | 3 months before treatment, 6 and 18 months after treatment has ended
  Montgomery Asberg Depression Rating Scale
Change from Baseline of obsessions and compulsions after 8 and 20 months. | 3 months before treatment, 6 and 18 months after treatment has ended
  Euroqol

CONTACTS AND LOCATIONS:
Locations (1):
- Psykiatri sydväst, Stockholm, Sweden

REFERENCES:
- See also: This is an amendment to NCT01347099 — http://clinicaltrials.gov